CLINICAL TRIAL: NCT07255950
Title: Accuracy Between Jabbing-then-suction, Suction-with-jabbing, and Suction-only Transthoracal Needle Aspiration (TTNA) Techniques in Suspected Lung Cancer Patients
Brief Title: Accuracy Between Transthoracal Needle Aspiration (TTNA) Techniques in Suspected Lung Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Siswanto Siswanto, Principal Investigator, Gadjah Mada University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KE/0943/06/2025
Record Dates: First submitted 2025-07-29; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer (Diagnosis); Biopsy, Fine-Needle/Methods
Keywords: NSCLC; Non-small cell lung cancer; Transthoracal needle aspiration; Biopsy; Diagnostics
MeSH Terms: conditions — Lung Neoplasms; Disease; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: All patient undergo the same intervention
Masking Description: The biopsy results, in a form of 20 cc syringe and slide containing the patient's tissue sample, will be labeled with a code by pulmonologist that will be blinded to the pathologist. The pathologist will then assess the adequacy of the cell count for molecular examination, evaluate the histopathological and cytopathological findings. Statisticians who will process the data are unaware of the allocation of each research item.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Jabbing-then-Suction, Suction-with-Jabbing, and Suction-only Transthoracal Needle Aspiration (TTNA) (Experimental)
  Interventions: Diagnostic Test: Jabbing-then-Suction, Suction-with-Jabbing, and Suction-only Transthoracal Needle Aspiration (TTNA) Techniques

INTERVENTIONS:
Diagnostic Test: Jabbing-then-Suction, Suction-with-Jabbing, and Suction-only Transthoracal Needle Aspiration (TTNA) Techniques — Each of patient will undergo three types of different transthoracal needle aspiration (TTNA)

SUMMARY:
* The objective of this research is to determine the accuracy of different types of lung transthoracal needle aspiration (TTNA) i.e. jabbing-then-suction, suction-with-jabbing, and suction-only TTNA in patients with suspected lung cancer.
* Researchers will compare these techniques to determine whether there are any quality differences in the obtained tumor samples

DETAILED DESCRIPTION:
During hospitalization for diagnostic testing, suspected lung cancer patients will undergo a transthoracic biopsy using three TTNA techniques, and core needle biopsy as the gold standard. The biopsy is performed in the operating room under local anesthesia and under the supervision of an anesthesiologist. The biopsy techniques used are routine procedures and therefore not as a new method. After the biopsy is completed, the patient is observed for at least 24 hours to observe potential complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected lung cancer who will undergo diagnostic testing using ultrasound-guided TTNA of the lung with cell block and core biopsy.
* Patients aged 18-75 years.
* The tumor is located peripherally, attached to the chest wall.

Exclusion Criteria:

* Patient refuses lung biopsy
* Non-cooperative patient
* Patient with respiratory failure, on positive pressure ventilation
* Severe pulmonary emphysema
* Contralateral pneumonectomy
* Advanced pulmonary fibrosis
* Platelet count <100,000/mm3 and international normalized ratio (INR) >1.4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Quality of samples from different types of transthoracal needle aspiration (TTNA) technique | Immediate after biopsy procedure
  To determine the quality of samples between the jabbing-then-suction technique, the suction-with-jabbing technique, and the suction-only technique of transthoracic needle aspiration procedures in patients with unsuspected lung cancer. The sample quality assessed includes the adequacy of the number of tumor cells for molecular examination and the concordance between cytology sample of each type of TTNA technique.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitas Gadjah Mada Academic Hospital (RSA UGM), Yogyakarta, Special Region of Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) collected during the trial reported in the article will be shared, after deidentification.
Supporting Information: Study Protocol
Time Frame: IPD and supporting information will be available immediately following publication, without end date.
Access Criteria: Requestors who provide a methodologically sound proposal can access the our IPD data. Proposals should be directed to roihan.iqbal@gmail.com